CLINICAL TRIAL: NCT02875756
Title: A Study Evaluating the Effect of the Number of Needle Revolutions Inside the Node on the Diagnostic Yield of EBUS-TBNA in Sarcoidosis
Brief Title: Effect of the Number of Needle Revolutions Inside the Node on the Diagnostic Yield of EBUS-TBNA in Sarcoidosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ritesh Agarwal, Additional Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NK/2232/study/1116
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 10 revolutions (Experimental): In this group, 10 revolutions will be made with the EBUS-TBNA needle
  Interventions: Procedure: 10 revolutions
- 20 revolutions (Active Comparator): In this group, 10 revolutions will be made with the EBUS-TBNA needle
  Interventions: Procedure: 20 revolutions

INTERVENTIONS:
Procedure: 10 revolutions — The 22G needle (Vizishot, Olympus) will be used to obtain specimens from the enlarged lymph nodes during EBUS. Once inside the lymph node, needle will be passed to and fro 10 times
  Arms: 10 revolutions
Procedure: 20 revolutions — The 22G needle (Vizishot, Olympus) will be used to obtain specimens from the enlarged lymph nodes during EBUS. Once inside the lymph node, needle will be passed to and fro 20 times
  Arms: 20 revolutions

SUMMARY:
The investigators plan to evaluate the effect of the number of needle revolutions inside the node on the diagnostic yield of endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) in patients with sarcoidosis.

DETAILED DESCRIPTION:
Sarcoidosis is a multisystem disorder of unknown etiology characterized by granulomatous inflammation involving various body organs. The diagnosis is made on the basis of compatible clinicoradiological feature, histopathologic evidence of non-caseating granuloma, and exclusion of other known causes for granulomatous inflammation. As the lung and mediastinal lymph nodes are the most commonly involved structures in sarcoidosis, various bronchoscopic techniques like endobronchial biopsy (EBB), transbronchial biopsy (TBLB) and transbronchial needle aspiration (TBNA) are needed for tissue sampling.

Among the bronchoscopic techniques, TBNA of lymph nodes has emerged as the most useful modality in addition to the previously known endobronchial and transbronchial biopsies. The efficacy and safety of conventional TBNA are well established. With improvements in technology, last decade has seen the use of EBUS to guide transbronchial needle aspiration. This technique is a minimally invasive and offers the additional advantage of choosing the appropriate node for sampling based on the vascularity, echogenicity and size. Studies subsequently have demonstrated the superiority EBUS-TBNA over conventional TBNA.

Once the role of TBNA in diagnostic bronchoscopy was clear, technical aspects of the procedure became the topic of research. This includes the number of aspirations or passes required per lymph node station, needle gauge (21 vs. 22 gauge), suction pressure, and the distance travelled by the needle within the lymph node. The number of revolutions i.e. the number of times the needle should be moved back-and-forth inside the lymph node is one such factor. The recommendation is to move the needle ten to twenty times. However the optimum number of times the needle should be moved back and forth for extracting adequate tissue material has not been studied to date. The investigators have observed that performing revolutions during EBUS-TBNA frequently leads to aspiration of blood during the procedure.

The investigators hypothesize that the number of revolutions will not affect the diagnostic yield, and the yield would be similar in 10 compared to 20 revolutions. In this study, the investigators plan to evaluate the effect of the number of needle revolutions inside the node on the diagnostic yield of EBUS-TBNA in patients with sarcoidosis.

ELIGIBILITY:
Inclusion Criteria:

* Age group of 18 to 65 years
* Clinicoradiological suspicion of sarcoidosis where EBUS-TBNA is being planned
* Enlarged hilar and mediastinal lymph nodes >10 mm (any axis) on computed tomography of the chest

Exclusion Criteria:

* Hypoxemia (SpO2 <92% on FiO2 of 0.3)
* Treatment with systemic glucocorticoids for >2 weeks in the preceding three months
* Diagnosis of sarcoidosis possible with another minimally invasive technique such as skin biopsy or peripheral lymph node biopsy
* Failure to provide informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-08; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield of EBUS-TBNA as indicated by the presence of granuloma | 1 week

SECONDARY OUTCOMES:
Adequacy of samples as indicated by the presence of lymphocytes | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Medical Education and Research, Chandigarh, Uttarakhand, India

IPD SHARING:
Plan to Share IPD: Undecided